CLINICAL TRIAL: NCT02543086
Title: A Phase1 Interventional Sequential Single Site Study to Characterize the Effectiveness of Oral KAE609 in Reducing Asexual & Sexual Blood-stage P. Falciparum Following Inoculation in Healthy-volunteers & Subsequent Infectivity to Mosquitoes
Brief Title: Effectiveness of KAE609 in Reducing Asexual & Sexual Blood-stage P.Falciparum Infection & Infectivity to Mosquitos
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Medicine for Malaria Venture (Unknown)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CKAE609A2109
Record Dates: First submitted 2015-07-23; First posted 2015-09-07 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: Phase 1, malaria, inoculum, P. falciparum, KAE609, Piperaquine
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — NITD 609; piperaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multiple Sequential Cohort (Experimental): This study is divided in 2 parts (Part A and part B). Each participant in each of the cohorts will be inoculated with viable parasites of Plasmodium falciparum-infected human erythrocytes administered intravenously. For Part A & Part B, commencement of treatment will be determined by Quantitative-Polymerase Chain Reaction results.
  The First cohort of Part A (A1) will be dosed with a single dose of KAE609. During Part A, an additional second single-dose of KAE609 may be tested (~15 days after first dose of KAE609 but may vary) if sexual parasitemia is identified. Subsequent cohorts of part A (An) will be dosed based on the results of first cohort (A1).
  Subjects enrolled in Cohort B will receive a pre-treatment with Piperaquine followed by KAE609 (~15 days).
  Interventions: Drug: KAE609; Drug: Piperaquine Phosphate

INTERVENTIONS:
Drug: KAE609 — Study drug
Drug: Piperaquine Phosphate — Pre-administration of Piperaquine Phosphate will be done to eliminate the asexual form of the parasite and induce gametocytaemia before characterizing the activity of KAE609 in clearing sexual blood stage parasites from the blood of healthy subjects in the Induced Blood Stage Malaria Challenge model in Part B of study

SUMMARY:
This is a single-center open label study conducted in multiple sequential cohorts using Induced Blood Stage Malaria infection in healthy volunteers to characterize the effectiveness of KAE609 against sexual and asexual blood stage forms of Plasmodium falciparum. This study is divided in 2 parts (Part A and part B). A total of 8 healthy volunteers per cohort will be enrolled. Based on the results of Part A, Part B will be undertaken to evaluate the effect of KAE609 following pretreatment with Piperaquine on sexual stage/gametocytemia and its activity as an inhibitor of onward transmission to mosquito vectors using experimental mosquito feeding assays.

DETAILED DESCRIPTION:
This is single center multiple sequential Cohort study divided in 2 parts (Part A and part B). A total of 8 healthy volunteers per cohort will be enrolled in Part A, which will focus on characterizing the antiparasitic activity of KAE609 after single dose administration in the human Induced Blood Stage Malaria model. Once Part A is completed, Part B will evaluate the effect of KAE609 following pre-treatment with Piperaquine on sexual stage/gametocytemia and its activity as an inhibitor of onward transmission to mosquito vectors using experimental mosquito feeding assays.

For Part A the threshold for commencement of treatment for an individual subject will occur if Quantitative-Polymerase Chain Reaction quantification of all participants in that Cohort is ≥ 1,000 parasites/mL or if Quantitative-Polymerase Chain Reaction quantification of any participant is ≥ 5,000 parasites/mL, and there is clinical evidence of malaria, as defined by a Clinical symptom score ≥6. The First cohort will be dosed with a single dose of KAE609. During Part A, an additional second single-dose of KAE609 for subsequent cohorts may be tested (~15 days after first dose of KAE609 but may vary) if sexual parasitemia is identified. Subsequent cohorts of part A (An) will be dosed based on the results of first cohort (A1).

For Part B, the threshold for commencement of treatment for an individual subject will be when Polymerase Chain Reaction quantification of all participants is ≥ 5,000 parasites/mL or if the Polymerase Chain Reaction quantification of any participant is ≥ 5,000 parasites/mL and is accompanied by a clinical symptom score ≥6, before all participants have reached the treatment threshold (PCR quantification of ≥ 5,000), then treatment of that participant will begin within a 24 h period. Cohort B will receive a pre-treatment with Piperaquine (480 mg) followed by KAE609 (~15 days) after Piperaquine.

Following initial treatment with KAE609 (Part A) or Piperaquine (Part B) on Day 1, participants will be followed up as in-subjects for at least 72 hours to ensure tolerance of the treatment and clinical response. If subjects are clinically well as per judgment of the Investigator, they will be discharged and will be monitored on an outpatient basis for safety and clearance of malaria parasites via Quantitative-Polymerase Chain Reaction. If any study subjects in a cohort in Part A show evidence of gametocytemia after initial treatment with KAE609, a second single-dose of KAE609 will be administered to those subjects as out patient. In part B where significant gametocytemia is expected because the initial Piperaquine treatment is not expected to clear gametocytes, a single dose of KAE609 will be administered at the time of peak gametocytemia. The KAE609 dose for Part B will be selected during the study, based on Pharmacokinetic/Pharmacodynamic and safety analysis of Part A. If recrudescent asexual parasitemia is identified, compulsory commencement of rescue medication will be used. Treatment for recrudescence will be a single dose of Piperaquine only for Part A. In addition, compulsory terminal curative treatment will be administered to all participants at the end of study. Participants will be monitored for three days to ensure adherence to the rescue medication therapy. Adverse events will be monitored via telephone monitoring, within the clinical research unit, and on out-subject review after malaria challenge inoculation and antimalarial study drug administration. Blood samples for safety evaluation, malaria monitoring, and red blood cell antibodies will be drawn at screening and/ or baseline and at nominated times after malaria challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any assessment is performed.
2. Male and females participants between 18 and 55 years of age. Female participants between 18 and 55 years of age have to be of non-child bearing potential.
3. Body weight, minimum 50.0 kg, body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.
4. Certified as healthy by a comprehensive clinical assessment.
5. Normal standard 12-lead electrocardiogram (ECG).
6. Laboratory parameters within the normal range.

Exclusion Criteria:

1. Any history of malaria or participation to a previous malaria challenge study
2. Spent more than four weeks in a malaria-endemic country during the past 12 months or planned travel to a malaria endemic area during the course of the study
3. Has evidence of increased cardiovascular disease risk
4. History of splenectomy
5. Presence or history of drug hypersensitivity, or allergic disease diagnosed
6. Presence of current or suspected serious chronic diseases
7. History of malignancy of any organ system
8. Presence of acute infectious disease or fever (e.g., sub-lingual temperature

   * 38.5°C) within the five days prior to inoculation with malaria parasites.
9. Participation in any investigational product study within the 12 weeks preceding the study.
10. Participant who has ever received a blood transfusion.
11. History or presence of alcohol abuse
12. Any vaccination within the last 28 days.
13. Any corticosteroids, anti-inflammatory drugs, immunomodulators or anticoagulants.
14. Any recent (< 1 month) or current systemic therapy with an antibiotic or drug with potential antimalarial activity (including chloroquine, piperaquine, tetracycline, azithromycin, clindamycin, hydroxychloroquine,).
15. Medicinal products that are known to prolong the QTc interval.
16. Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, antihepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti HIV2 Ab).
17. Known severe reaction to mosquito bites other than local itching and redness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-07; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Parasitic count in blood by Polymerase Chain Reaction | 36 days
  Clearance of Plasmodium falciparum asexual and sexual blood stage parasites from the blood of healthy subjects in the Induced Blood Stage Malaria Challenge model

SECONDARY OUTCOMES:
Plasma Pharmacokinetics (PK) of KAE609: Area Under the Plasma Concentration-time Curve (AUC) | Day 1: 0, 1, 2, 3, 4, 8, 12, 16 hours, then 24, 36, 48, 72, 96 and 120 hours post dose Days 2 to 6, Day 15 0, 12 hours post dose then 24, 48, 72, 96 and 120 hours post dose Day 16 to Day 20
  It will be measured by Area Under the Concentration-Time Curve (AUC) from the time of dosing to the last quantifiable concentration
Safety and Tolerability as measured by adverse events (including serious) for incidence, KAE609 (and inoculum) relatedness and severity | From day of screening until end of study (day 36)
  Adverse events (including serious) will be recorded during the study and will be rated according to incidence, relation to study drug (inoculum) and severity

CONTACTS AND LOCATIONS:
Overall Officials: James McCarthy, MD FRACP, Principal Investigator — Q-Pharm Pty Limited
Locations (1):
- Novartis Investigative Site, Brisbane, Queensland, Australia

REFERENCES:
- [Derived] McCarthy JS, Abd-Rahman AN, Collins KA, Marquart L, Griffin P, Kummel A, Fuchs A, Winnips C, Mishra V, Csermak-Renner K, Jain JP, Gandhi P. Defining the Antimalarial Activity of Cipargamin in Healthy Volunteers Experimentally Infected with Blood-Stage Plasmodium falciparum. Antimicrob Agents Chemother. 2021 Jan 20;65(2):e01423-20. doi: 10.1128/AAC.01423-20. Print 2021 Jan 20. PMID 33199389